CLINICAL TRIAL: NCT01724203
Title: Effect of 12-week Probiotic Supplementation on Bacterial and Viral Infections in Infants Aged 6 to 12 Months: a Double-blind, Randomized, Placebo-controlled Study.
Brief Title: Effect of 12-week Probiotic Supplementation on Bacterial and Viral Infections in Infants Aged 6 to 12 Months.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fonterra Research Centre (Industry)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 111104-SUS-FON-ICP-MS
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Effect of Probiotics on Infections in Infants.
Keywords: Probiotics for infants; Bacterial and viral infections in infants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lactobacillus rhamnosus (Active Comparator): Formula containing 1 million CFU/g Lactobacillus rhamnosus HN001 (trademarked DR20) at least three times daily for 12 weeks.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus
- Bifidobacterium animalis subsp. lactis (Active Comparator): Formula containing 1 million CFU/g Bifidobacterium animalis subsp. lactis HN019 (trademarked DR10) at least three times daily for 12 weeks.
  Interventions: Dietary Supplement: Bifidobacterium animalis subsp. lactis
- Placebo (Placebo Comparator): Placebo formula without probiotics at least three times daily for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus
  Arms: Lactobacillus rhamnosus
Dietary Supplement: Bifidobacterium animalis subsp. lactis
  Arms: Bifidobacterium animalis subsp. lactis
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and effectiveness of 12-week probiotic supplementation on the incidence and duration of infectious episodes in infants aged 6 to 12 months.

DETAILED DESCRIPTION:
Probiotics are live bacteria that offer a health benefit to the host when administered via the diet in adequate amounts. Probiotic supplementation is safe for use in infants to the elderly and has demonstrated beneficial effects for a wide variety of health conditions such as acute diarrhea, antibiotic-associated diarrhea, allergies, and inflammatory bowel disease. The immune-enhancing benefits of probiotics are attractive, particularly for infants, a group that is particularly prone to a variety of infections, e.g. respiratory tract infection, strep throat, and diarrhea. Probiotic supplementation has been utilized in previous studies of childhood infections with promising results.

In this study, the safety and effectiveness of 12-week probiotic supplementation on the incidence and duration of infectious episodes in infants aged 6 to 12 months will be determined. The subjects will receive follow-on formula containing 1 million CFU/g Lactobacillus rhamnosus HN001 (trademarked DR20), 1 million CFU/g Bifidobacterium animalis subsp. lactis HN019 (trademarked DR10), or placebo formula for at least three feeds per day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 months.
* Known vaccination history.
* Ability of the participant's parent or legal guardian to comprehend the full nature and purpose of the study including possible risks and side effects.
* Parental or legal guardian's consent to the study and willing to comply with study procedures.

Exclusion Criteria:

* Symptoms of any infection at screening.
* History of ≥5 infections in the previous 2 months.
* Lactose intolerance or unable to drink milk.
* Leukopenia or leukocytosis.
* Immunodeficient or use of immunosuppressive drugs.
* Use of antibiotic and anti-inflammatory medications within the last 2 weeks.
* Use of products containing prebiotics or probiotics within the last 2 weeks.
* Use of low-lactose or lactose-free infant or follow-on formula within the last 2 weeks.
* Hepatitis B or C.
* Medications or supplements that may affect subject safety or confound study outcomes in the opinion of the investigator.
* Medical conditions or diseases that may affect subject safety or confound study results in the opinion of the investigator.
* Participation in another study with any investigational product within 3 months of screening.
* Any other condition that, in the investigator's opinion, may preclude the subject's ability to safely complete the trial.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with one or more of confirmed bacterial or viral infections at any time during the study | 12 weeks
  The primary endpoint of this clinical trial is the proportion of subjects with one or more of the following confirmed bacterial or viral infections at any time during the study: fever > 37.5ºC (axillary), upper respiratory tract infection, lower respiratory tract infection, pneumonia, strep throat, diarrhea, and otitis media.

SECONDARY OUTCOMES:
Cumulative days with infectious symptoms | 12 weeks
  Cumulative number of days with infectious symptoms will be defined as the total number of days during the study on which a subject has symptoms of a confirmed infection. Confirmed infections that count toward the primary endpoint include: fever >37.5°C (axillary), upper respiratory tract infection, lower respiratory tract infection, pneumonia, strep throat, diarrhea, and otitis media.
Cumulative number of infectious episodes | 12 weeks
  Cumulative number of infectious episodes will be defined as the total number of infectious episodes (defined as presence of one of more symptoms of a confirmed infection) experienced during the study. An infectious episode will be defined as a period when symptoms of a confirmed infection last for more than 24 hours and are followed by at least 3 days of no symptoms.
Stool frequency | 12 weeks
  Parents will record the number of infant defecations each day in a diary during the 12-week supplementation period.
Stool Consistency | 12 weeks
  Parents will rate the consistency of each infant bowel movement by using the Bristol Stool Scale Form. Parents will record stool consistency each day during the 12-week supplementation period.
Infant Characteristics Questionnaire | 12 weeks
  The Infant Characteristic Questionnaire for infants approximately 6 months old (ICQ-6) measures parental perception of infant temperament, focusing on difficult temperament 8. The questionnaire is comprised of 24 items describing infant behavior. The parent or primary caregiver ranks each item on a 7-point scale, indicating the level of perceived difficulty in dealing with the described behavior. Four subscales have been identified through principal components analyses: Fussy/Difficult, Unadaptable, Dull, and Unpredictable.
Treatments for infectious episodes | 12 weeks
  Treatments that are taken to alleviate infectious symptoms will be documented in a daily diary.
Adverse events | 12 weeks
  Adverse events will be recorded in the daily diary and at study visits during the 12-week supplementation period.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Sheng, Dr, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Dekker J, Quilter M, Qian H. Comparison of two probiotics in follow-on formula: Bifidobacterium animalis subsp. lactis HN019 reduced upper respiratory tract infections in Chinese infants. Benef Microbes. 2022 Oct 4;13(4):341-354. doi: 10.3920/BM2022.0041. Epub 2022 Aug 25. PMID 36004715